CLINICAL TRIAL: NCT04081675
Title: Understanding the Factors Affecting Compliance in Children With Cerebral Palsy Supplied With Ankle Foot Orthoses (AFOs) Using Quantitative Measurement of Function and Qualitative Evaluation of Experience and Wellbeing
Brief Title: Compliance in Children With Cerebral Palsy Supplied With AFOs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Keele University (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: RL1796
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy
Keywords: orthotics; gait analysis
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ankle Foot Orthosis (AFO) — Thermoplastic orthotic device spanning the calf, ankle and foot.

SUMMARY:
Children with cerebral palsy are frequently supplied with Ankle Foot Orthoses (AFOs) to aid their walking. There are huge benefits to patients in staying physically active into adulthood but this becomes more challenging as children progress through adolescence. It is possible to measure the functional benefits of AFO use, however the investigators suspect the correlation with patient compliance is poor. By combining quantitative analysis using 3D gait analysis with qualitative exploration of children's experience the investigators hope to gain a better understanding of the factors influencing children's compliance. This compliance will be measured using sensors mounted in the AFOs, over a 3 month period. The investigators hope this research will help clinicians manage patients better and also inform changes in splint design.

DETAILED DESCRIPTION:
Background

About 1 in 400 children born in the UK has cerebral palsy (CP). CP is caused by injury to the foetal or infant brain, and results in problems with walking, balance and coordination. One of the most common strategies for treating walking limitations in children with CP is the use of Ankle Foot Orthoses (AFOs), which aim to correct deformity and improve walking efficiency.

Keeping children with CP mobile is important, not only because physical fitness contributes to quality of life, but also because lack of physical activity can result in a downwards spiral: low physical fitness can make activities of daily living more difficult, leading to further reduction in activity and fitness. One study showed that children with CP at age 10 who walked and did not use a wheelchair had only a small chance (11%) of becoming non-ambulatory, vs. 34% of children using a wheelchair.

AFOs can play an important part in keeping children with CP mobile, and reducing the need for a wheelchair. However, there is evidence that when they reach adolescence, some children are reluctant to wear their AFOs. One of the parents participating in a previous study said "... now we have a 13-year-old who just wants to be like other 13- year-old girls, and she doesn't want to wear AFOs ...". Studies show that children with CP often lose functional ability through adolescence and early adulthood, but it is not clear how that relates to their use or non-use of prescribed AFOs. There are also many factors which contribute to compliance with clinical recommendation and a scarcity of research into the psychological elements which can impact on this, though research indicates that perception and empowerment can increase the likelihood of a successful intervention application and compliance rates.

In this application the investigators seek to explore both the objective, functional benefits of using AFOs and the subjective experience of children and their families. A combination of quantitative and qualitative approaches will be used to understand the factors affecting children's compliance.

Purpose, aims or hypothesis

The overall aim is to understand the factors affecting compliance in children with cerebral palsy using AFOs. The investigators propose to do this by combining quantitative measurement of functional benefit, with qualitative exploration of the patient's experience.

To achieve this the investigators will:- Phase 1: Measure the functional effect of AFOs using 3D movement analysis technology in four children (treated as case studies).

Phase 2: Record patient compliance in the same group of children using sensors embedded in the AFOs Phase 3: Interview children and their families to explore the experience of using assistive devices.

Experimental plan, methods, timetable:

Children with cerebral palsy will be recruited from the routine clinics in ORLAU, at the RJAH Orthopaedic Hospital. The investigators will aim to recruit 4 children with cerebral palsy who have been prescribed bilateral moulded AFOs, two from primary school years 5/6 (1F, 1M) and two from secondary school years 7-9 (1F, 1M). The children will be GMFCS level 1 or 2 and be in main stream education.

Phase 1: 3D movement analysis

Children will be measured by means of 3D movement analysis (Vicon) at their supply appointment. Markers will be placed on the lower limbs and pelvis using the Plug-in-Gait model. Children will be measured walking in shoes with and without their AFOs. The gait analysis will provide detailed quantification of angles and moments at each joint, however the primary measures will be walking speed and the collated GPS which gives an overall score of the deviation from normal walking.

A full clinical examination will also be performed, along with video film of their feet when walking barefoot to assess the extent of any foot deformity.

Phase 2: Assessment of compliance

Each AFO will be fitted with an Orthotimer (www.orthotimer.com) sensor before it is supplied. This data will be downloaded at the review appointment, when the interviews will also be conducted. The device stores data every 15 min for up to 100 days recording whether the orthosis is in use at a given time.

Phase 3: Interviews

Semi-structured interviews will take place with the children recruited for phase 1, asking questions which will allow them to discuss their experiences of living with CP and of using assistive devices, particularly within their school environment; participants in secondary school will be also be asked about their experience in primary school. Questions will be as open as possible to allow the child to give rich, detailed accounts of their day to day experiences and their perceptions of AFOs. The interviews should provide a broad understanding of individual experiences and perspectives of AFOs and reasons for compliance. All children and their families will be invited back to verify the themes from the interviews at a separate, non-clinical, visit. Themes from the school group sessions will be used to shape the questions.

A mapping exercise, based on previous research will be used to enhance the discussion and visually identify locations where the children use their AFOs, their feelings triggered by a range of environments, and any issues they may have with the orthotic devices. These maps can then be used to facilitate further discussion about the children's experiences and analysed alongside the Orthotimer data to develop an in-depth view of the children's use and perception of their AFOs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic diplegia or hemiplegia GMFCS level 1 or 2 (ie independently mobile) Gait pattern compatible with achieving clean foot strikes on the force platforms in the gait laboratory.
* Able to understand sufficiently to co-operate happily with the gait analysis process and participate in the interviews.
* In main stream education

Exclusion Criteria:

* Any behavioural or communication problems which would make them unable to comply with the protocol.
* Any invasive procedures (eg surgery, Botulinum toxin injections) in the previous 6 months.
* Any invasive procedures (eg surgery, Botulinum toxin injections) planned in the next 6 months.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Walking speed (m/s) | At baseline
  This will be measured in a clinical movement analysis laboratory using timing gates at either end of the walkway.
Gait Profile Score (GPS) in degrees | At baseline
  A 3D movement analysis system will be used to record the full kinematics and kinetics of the child's gait with and without AFOs. The outcome measure extracted will be the GPS, which documents the average deviation in joint angles (in degrees) across multiple joints compared with an unimpaired control cohort. Unimpaired data are already available in the host unit.
Compliance (minutes per day) | At end of 3 months of use
  The compliance will be recorded using Orthotimer sensors embedded in the body of the AFO. The sensors record usage throughout the day in 15min intervals.
Patient Experience | At end of 3 months of use
  Qualitative interviews - an entirely qualitative approach will be used to draw out narrative themes. No scoring scale is used.

CONTACTS AND LOCATIONS:
Overall Officials: Dr C Stewart, PhD, Principal Investigator — RJAH Orthopaedic Hospital/Keele University
Locations (1):
- ORLAU, RJAH Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson C, Mattsson E. Adults with cerebral palsy: a survey describing problems, needs, and resources, with special emphasis on locomotion. Dev Med Child Neurol. 2001 Feb;43(2):76-82. doi: 10.1017/s0012162201. PMID 11221908
- [Background] Butler PB, Farmer SE, Stewart C, Jones PW, Forward M. The effect of fixed ankle foot orthoses in children with cerebral palsy. Disabil Rehabil Assist Technol. 2007 Jan;2(1):51-8. doi: 10.1080/17483100600662009. PMID 19263554
- [Background] Day SM, Wu YW, Strauss DJ, Shavelle RM, Reynolds RJ. Change in ambulatory ability of adolescents and young adults with cerebral palsy. Dev Med Child Neurol. 2007 Sep;49(9):647-53. doi: 10.1111/j.1469-8749.2007.00647.x. PMID 17718819
- [Background] Gabb J, Singh R. The uses of emotion maps in research and clinical practice with families and couples: methodological innovation and critical inquiry. Fam Process. 2015 Mar;54(1):185-97. doi: 10.1111/famp.12096. Epub 2014 Aug 5. PMID 25091031
- [Background] Hayles E, Harvey D, Plummer D, Jones A. Parents' Experiences of Health Care for Their Children With Cerebral Palsy. Qual Health Res. 2015 Aug;25(8):1139-54. doi: 10.1177/1049732315570122. Epub 2015 Feb 23. PMID 25711842
- [Background] Prevalence and characteristics of children with cerebral palsy in Europe. Dev Med Child Neurol. 2002 Sep;44(9):633-40. PMID 12227618
- [Background] Koldoff EA, Holtzclaw BJ. Physical Activity Among Adolescents with Cerebral Palsy: An Integrative Review. J Pediatr Nurs. 2015 Sep-Oct;30(5):e105-17. doi: 10.1016/j.pedn.2015.05.027. Epub 2015 Jul 18. PMID 26195302
- [Background] Krakovsky G, Huth MM, Lin L, Levin RS. Functional changes in children, adolescents, and young adults with cerebral palsy. Res Dev Disabil. 2007 Jul-Sep;28(4):331-40. doi: 10.1016/j.ridd.2006.03.005. PMID 16772110
- [Background] Nooijen C, Slaman J, van der Slot W, Stam H, Roebroeck M, van den Berg-Emons R; Learn2Move Research Group. Health-related physical fitness of ambulatory adolescents and young adults with spastic cerebral palsy. J Rehabil Med. 2014 Jul;46(7):642-7. doi: 10.2340/16501977-1821. PMID 24714702
- [Background] Wingstrand M, Hagglund G, Rodby-Bousquet E. Ankle-foot orthoses in children with cerebral palsy: a cross sectional population based study of 2200 children. BMC Musculoskelet Disord. 2014 Oct 2;15:327. doi: 10.1186/1471-2474-15-327. PMID 25274143